CLINICAL TRIAL: NCT06202612
Title: A Bioavailability Study of SHR0302 Tablet in Healthy Subjects
Brief Title: A SHR0302 BA Study on Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR0302-113
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: There will be two independent cohorts of subjects who will each receive two treatments (quick release tablets and sustained-release tablets), and each treatment will be followed by 72 hours of blood sampling for pharmacokinetic assessments, with safety and tolerability.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR0302 quick release tablet and sustained-release tablet (Experimental)
  Interventions: Drug: SHR0302 quick release tablets; Drug: SHR0302 sustained-release tablets
- SHR0302 sustained-release tablet and quick release tablet (Experimental)
  Interventions: Drug: SHR0302 quick release tablets; Drug: SHR0302 sustained-release tablets

INTERVENTIONS:
Drug: SHR0302 quick release tablets — SHR0302 quick release tablets 8 mg
Drug: SHR0302 sustained-release tablets — SHR0302 sustained-release tablets 10 mg

SUMMARY:
The purpose of this study is to evaluate and compare the pharmacokinetics of SHR0302 two different kind tablets in Healthy subjects after administration two kind tablets (quick release tablets and sustained-release tablets).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy subjects aged 18 to 60 (including 18 and 60);
2. Weigh at least 50 kg (for male) and 45 kg (for female), respectively, and have a body mass index (BMI) ≥ 19 and ≤26 kg/m2. BMI = weight (kg)/[height (m)]2;
3. From the signing of the informed consent form until 6 months after the last administration, the subject (including partner) has no family planning and is willing to use the high-efficiency contraceptive measures specified in the plan;
4. Sign the informed consent before the trial, and fully understand the content, process and possible adverse reactions of the trial. Must be able to communicate with the investigator, understand and comply with all study requirements.

Exclusion Criteria:

1. Any clinical history of serious diseases or conditions that the researcher believes may affect the trial results, including but not limited to circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic disease history;
2. Those who have a history of tuberculosis within 6 months before signing the informed consent form; Or those who tested positive for T-spot test within the first 4 weeks of randomization;
3. Individuals who have a history of smoking (average daily smoking>5 cigarettes) within the 3 months prior to signing the informed consent form, or who cannot stop using any tobacco products during the study period;
4. Those who consume more than 25 g of alcohol per day on average within three months before signing the informed consent form (for example, 750 mL of beer, 250 mL of wine, or 50 mL of Baijiu), or cannot stop using any alcoholic products during the study period, or those who are positive in the alcohol breath test during screening;
5. Drug abusers, or those who have tested positive for urinary drug abuse during screening, including: morphine, methamphetamine, ketamine, cocaine, ecstasy (dimethylenedioxoamphetamine), marijuana (tetrahydrocannabidiol acid);
6. During the screening period, if the QTc of the ECG examination is greater than 450 ms or there are other clinically significant abnormalities determined by the researcher;
7. Vital signs, physical examinations, laboratory tests, abdominal ultrasound or chest imaging examinations during the screening period indicate the presence of abnormalities that have been determined by the researchers to be clinically significant;
8. Hepatitis B surface antigen (HBsAg) positive, or anti hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody positive, or syphilis antibody positive;
9. Within the first 7 days of randomization, any beverage or food containing grapefruit, grapefruit, strong tea, coffee, mangoes, etc. was consumed;
10. Allergic constitution, or suspected allergy to any component of SHR0302 medication;
11. Infections that require systemic antimicrobial therapy that occurred within the first 4 weeks of randomization (viral, bacterial, fungal, parasitic infections);
12. Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or dietary supplements within the first two weeks of randomization;
13. Systemic treatment with inhibitors or inducers of cytochrome P450 3A4 enzyme (CYP3A4) within the first 4 weeks of randomization (see Annex 2 for details);
14. Individuals who participated in any drug clinical trial and took the investigational drug within the first three months of randomization (calculated from the last visit of the previous trial) (if the five half-lives of the investigational drug exceed three months, the time of the five half-lives shall prevail);
15. Received BCG vaccine within the first 12 months of randomization; Or receive or be exposed to other live vaccines or attenuated live vaccines within the first three months of randomization; Or those who plan to receive the vaccine during the trial period;
16. Individuals who have undergone any surgery within the first three months of randomization, or who have not yet recovered after surgery, or who are expected to have surgery or hospitalization plans during the trial period;
17. Individuals who have donated (or lost) blood within the first three months of randomization and have donated (or lost) ≥ 400 mL of blood, or have received blood transfusions;
18. According to the researcher's judgment, the subjects may have factors that affect drug absorption, distribution, metabolism, and excretion, or other factors that are not suitable for participation in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
PK parameters of SHR0302: Cmax | Based on pre-dose, 0.25-72 hours post-dose sampling times after administration on Day 1 and Day 5
PK parameters of SHR0302: AUC0-t | Based on pre-dose, 0.25-72 hours post-dose sampling times after administration on Day1 and Day 5
PK parameters of SHR0302: AUC0-inf | Based on pre-dose, 0.25-72 hours post-dose sampling times after administration on Day 1 and Day 5
Relative bioavailability (F%) between SHR0302 sustained-release tablets and SHR0302 rapid release tablets | Based on pre-dose, 0.25-72 hours post-dose sampling times after administration on Day 1 and Day 5
  F%=AUC (sustained-release tablets) * dose (rapid release tablets)/AUC (rapid release tablets) * dose (sustained-release tablets) × 100%

SECONDARY OUTCOMES:
PK parameters of SHR0302: Tmax | 0 hour to 72 hour after administration with sustained-release tablets or rapid release tablets on Day 1 and Day 5
PK parameters of SHR0302: t1/2 | 0 hour to 72 hour after administration with sustained-release tablets or rapid release tablets on Day 1 and Day 5
PK parameters of SHR0302: CL/F | 0 hour to 72 hour after administration with sustained-release tablets or rapid release tablets on Day 1 and Day 5
PK parameters of SHR0302: Vz/F | 0 hour to 72 hour after administration with sustained-release tablets or rapid release tablets on Day 1 and Day 5
Adverse events of SHR0302 with sustained-release tablets or rapid release tablets | from ICF signing date to day 12 (±1)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided